CLINICAL TRIAL: NCT05785832
Title: A Randomized Trial Evaluating the Efficacy and Safety of Control-IQ+ Technology in Adults With Type 2 Diabetes Using Basal-Bolus Insulin Therapy (2IQP)
Brief Title: A Randomized Trial Evaluating Control-IQ+ Technology in Adults With Type 2 Diabetes
Acronym: 2IQP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP-0013437
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: Control-IQ+ technology; type 2 diabetes; automated insulin dosing; automated insulin delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Intervention group (Experimental): t:slim X2 insulin pump with Control-IQ+ technology and Dexcom G6 CGM for 13 weeks.
  Interventions: Device: t:slim X2 insulin pump with Control-IQ+ technology and Dexcom G6 CGM
- Control group (Active Comparator): Continuation of pre-study basal-bolus insulin delivery method, plus use of study CGM (Dexcom G6) for 13 weeks.
  Interventions: Device: Standard Therapy plus continuous glucose monitoring (CGM)

INTERVENTIONS:
Device: t:slim X2 insulin pump with Control-IQ+ technology and Dexcom G6 CGM — The t:slim X2 insulin pump with Control-IQ+ technology, used with the Dexcom G6 CGM.
  Arms: Intervention group
Device: Standard Therapy plus continuous glucose monitoring (CGM) — Standard therapy is continuation of pre-study basal-bolus insulin delivery method, plus use of Dexcom G6 CGM.
  Arms: Control group

SUMMARY:
A randomized controlled trial (RCT) to assess the safety and efficacy of use of Control-IQ+ technology in adults with type 2 diabetes using basal-bolus insulin therapy.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) will evaluate 13 weeks of home use of the t:slim X2 insulin pump with Control-IQ+ technology in adults with type 2 diabetes age 18 and older using basal-bolus insulin therapy compared with continuation of pre-study insulin delivery plus continuous glucose monitoring (CGM). At least 300 participants will complete the trial at up to 25 clinical sites, across the United States and Canada.

Participants who skip or successfully complete the run-in will be randomly assigned 2:1 to the intervention group using the t:slim X2 insulin pump with Control-IQ+ technology or to continue their pretrial insulin-delivery method for 13 weeks. Both arms used the Dexcom G6 CGM.

The primary outcome is change in hemoglobin A1c (HbA1c) compared between the intervention and control group. The secondary endpoints will be tested for superiority, with a hierarchical testing approach. Additional outcomes are exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old at time of screening.
* Currently resides in the U.S. or Canada with the ability to complete in-person study visits at one of the participating clinical sites.
* Clinical diagnosis, based on investigator assessment, of type 2 diabetes of at least 6 months duration at time of screening.
* Using basal-bolus insulin therapy with at least one injection containing rapid-acting insulin per day or an insulin pump for at least 3 months prior to enrollment, with no major modification to insulin regime in the last 3 months (mixed insulin with a rapid component is acceptable).
* If using noninsulin glucose-lowering medications (such as GLP-1 receptor agonist, SGLT2 inhibitor, or other) or weight-reduction medications, dose has been stable for the 3 months prior to screening; and participant is willing to not change the dose unless required for safety purposes.
* Participant willing to not initiate use of any new glucose-lowering medications during the trial.
* Willing to use an approved insulin while using the study pump if assigned to the AID group.
* Willing to not use concentrated insulin above U-100 or inhaled insulin while using the study pump.
* Willing to participate in the study meal and exercise challenges if assigned to the AID group, and have a care partner, trained in hypoglycemia treatment guidelines, to include glucagon use, present during and immediately after the exercise challenges.
* Has the ability to read and understand written English.
* Investigator believes that the participant has the cognitive capacity to provide informed consent.
* Investigator believes that the participant can successfully and safely operate all study devices and is capable of adhering to the protocol and completing the study.
* No medical, psychiatric, or other conditions, or medications being taken that in the investigator's judgement would be a safety concern for participation in the study. This includes considering the potential impact of medical conditions known to be present including cardiovascular, liver, kidney disease, thyroid disease, adrenal disease, malignancies, vision difficulties, active proliferative retinopathy, and other medical conditions; psychiatric conditions including eating disorders; drug or alcohol abuse.
* Participants capable of becoming pregnant must meet one of the following criteria:

  1. has a negative urine pregnancy test and agrees to use one of the accepted contraceptive regimens throughout the entire duration of the trial from screening until last follow-up visit. The following contraceptive measures are considered adequate:

     1. Combined estrogen and progestogen containing hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal).
     2. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable).
     3. Placement of an intrauterine device or intrauterine hormone-releasing system.
     4. Bilateral tubal occlusion.
     5. Barrier methods of contraception (condom or occlusive cap with spermicidal foam/gel/film/cream/suppository).
     6. Has a vasectomized or sterile partner (where partner is sole partner of subject) and where vasectomy has been confirmed by medical assessment.
     7. Exercises true sexual abstinence. Sexual abstinence is defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.

     or
  2. Participant is of non-childbearing potential due to menopause with at least one year since last menses or a medical condition confirmed by the investigator.

Exclusion Criteria:

* Current use of hybrid closed-loop system.
* Current use of systemic glucocorticoids or anticipated use of glucocorticoids during the RCT (topical or inhaled -ie, non-systemic is acceptable).
* Current use of sulfonylurea or meglitinide medications.
* Current use of hydroxyurea.
* Tape allergy or skin condition that will preclude use of the study pump or CGM.
* Presence of a hemoglobinopathy or other condition that is expected to affect the measurement of HbA1c.
* Pregnant (positive urine hCG), breast feeding, plan to become pregnant in the next 2 months, or sexually active without use of contraception.
* Current participation in another diabetes-related interventional clinical trial.
* Anticipated change of residency or travel for more than 7 days at a time during the study that may, per investigator judgment, interfere with the completion of study visits, contacts, or procedures.
* Immediate family member (spouse, biological or legal guardian, child, sibling, parent) who is an investigative site personnel directly affiliated with this study or who is an employee of Tandem Diabetes Care, Inc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Pinsker, MD, Study Director — Tandem Diabetes Care; Yogish Kudva, MBBS, Study Chair — Mayo Clinic
Locations (21):
- United States (19):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - Baltimore VA Medical Center, Baltimore, Maryland
  - Boston Medical Center Corporation, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - UHH Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Diabetes and Endocrinology, P.A., Austin, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Diabetes & Endocrine Treatment Specialists, Sandy City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Rainier Clinical Research Center, Renton, Washington
  - University of Washington, Seattle, Washington
- Canada (2):
  - Lawson Health Research Institute, London, Ontario
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kudva YC, Raghinaru D, Lum JW, Graham TE, Liljenquist D, Spanakis EK, Pasquel FJ, Ahmann A, Ahn DT, Aleppo G, Blevins T, Kruger D, Brown SA, Levy CJ, Weinstock RS, Steenkamp DW, Spaic T, Hirsch IB, Broyles F, Rickels MR, Tsoukas MA, Raskin P, Hatipoglu B, Desjardins D, Terry AN, Singh LG, Davis GM, Schmid C, Kravarusic J, Coyne K, Casaubon L, Espinosa V, Jones JK, Estrada K, Afreen S, Levister C, O'Malley G, Liu SL, Marks S, Peleckis AJ, Pasqua MR, Tardio V, Kurek C, Luker RD, Churchill J, Tajrishi FZ, Dean A, Dennis B, Fronczyk E, Perez J, Mukhashen S, Dhillon J, Ipek A, Bzdick S, Atakov Castillo A, Driscoll M, Averkiou X, Dalton-Bakes CV, Moore A, Jordan LF, Lesniak A, Pinsker JE, Sasson-Katchalski R, Campos T, Spanbauer C, Kanapka L, Kollman C, Beck RW; 2IQP Study Group. A Randomized Trial of Automated Insulin Delivery in Type 2 Diabetes. N Engl J Med. 2025 May 8;392(18):1801-1812. doi: 10.1056/NEJMoa2415948. Epub 2025 Mar 19. PMID 40105270
- [Result] Hirsch IB, Kudva YC, Ahn DT, Blevins T, Rickels MR, Raghinaru D, Lum JW, Kollman C, Pinsker JE, Beck RW; 2IQP Study Group*. Adults With Type 2 Diabetes Benefit From Automated Insulin Delivery Irrespective of C-Peptide Level. Diabetes Care. 2025 Dec 1;48(12):2061-2066. doi: 10.2337/dc25-1125. PMID 40953318

RESULTS

PARTICIPANT FLOW:
Groups:
- Control-IQ+ AID: t:slim X2 insulin pump with Control-IQ+ technology and Dexcom G6 CGM for 13 weeks.
- CGM Arm: Continuation of pre-study basal-bolus insulin delivery method, plus use of study CGM (Dexcom G6) for 13 weeks.
Period: Overall Study
Arm/Group | Control-IQ+ AID | CGM Arm
Started | 215 | 104
Completed | 211 | 102
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control-IQ+ AID | CGM Arm | Total
Number analyzed (Participants) | 215 | 104 | 319
Age, Continuous [Mean (Standard Deviation); unit: year] | 59 (12) | 57 (12) | 57 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 49 | 154
  Male | 110 | 55 | 165
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 10 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 45 | 24 | 69
  White | 148 | 74 | 222
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 14 | 6 | 20
  United States | 201 | 98 | 299

OUTCOME MEASURES:

1. Primary Outcome: HbA1c
Description: Change in HbA1c (%) from baseline between the intervention and control groups
Time Frame: 13 weeks
Population: Data were missing because the sample that was obtained from one patient could not be analyzed.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 214 | 104
percentage of glycated hemoglobin
  Baseline | 8.2 (1.4) | 8.1 (1.2)
  13 Weeks | 7.3 (0.9) | 7.7 (1.1)
  Change from Baseline | -0.9 (1.1) | -0.3 (0.9)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -0.6, 95% CI 2-sided [-0.8 to -0.4]

2. Secondary Outcome: Time in Range 70-180 mg/dL
Description: Change in CGM percent time 70-180 mg/dL from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
percentage of time
  Baseline | 48 (24) | 51 (21)
  13 Weeks | 64 (16) | 52 (21)
  Change from Baseline | 16 (19) | 1 (14)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = 14, 95% CI 2-sided [11 to 17]

3. Secondary Outcome: Mean Glucose
Description: Change in mean CGM glucose mg/dL from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
mg/dL
  Baseline | 194 (43) | 190 (35)
  13 Weeks | 170 (23) | 188 (34)
  Change from Baseline | -24 (34) | -1 (24)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -21, 95% CI 2-sided [-26 to -15]

4. Secondary Outcome: Time >180 mg/dL
Description: Change in CGM percent time >180 mg/dL from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
percentage of time
  Baseline | 51 (25) | 49 (21)
  13 Weeks | 35 (16) | 48 (21)
  Change from Baseline | -16 (19) | -1 (14)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -14, 95% CI 2-sided [-17 to -11]

5. Secondary Outcome: Time >250 mg/dL
Description: Change in CGM percent time >250 mg/dL from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
percentage of time
  Baseline | 19.5 (17.3) | 15.8 (13.6)
  13 Weeks | 9.7 (7.8) | 16.7 (14.1)
  Change from Baseline | -9.7 (17.1) | 1.0 (11.4)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -9.1, 95% CI 2-sided [-11.7 to -6.6]

6. Secondary Outcome: Prolonged Hyperglycemia Events Per Week
Description: Change in number of prolonged hyperglycemia events (>90 minutes >300 mg/dL within a 120-minute period) per week from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: events per week
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
events per week
  Baseline | 1.7 (1.7) | 1.6 (1.7)
  13 Weeks | 0.9 (0.9) | 1.6 (1.5)
  Change from Baseline | -0.7 (1.5) | 0.0 (1.0)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.0 to -0.4]

7. Secondary Outcome: Time <70 mg/dL
Description: Change in CGM percent time <70 mg/dL from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
percentage of time
  Baseline | 0.7 (0.8) | 0.3 (0.3)
  13 Weeks | 0.4 (0.4) | 0.4 (0.4)
  Change from Baseline | -0.2 (1.2) | 0.1 (0.6)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Regression, Linear — A hierarchical procedure was used to control for the overall type I error. Since the P value for this outcome was more than 0.05, no additional P values are provided for subsequent secondary outcomes; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.1]

8. Secondary Outcome: Time <54 mg/dL
Description: Change in CGM percent time <54 mg/dL from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
percentage of time
  Baseline | 0.16 (0.16) | 0.05 (0.05)
  13 Weeks | 0.09 (0.09) | 0.09 (0.10)
  Change from Baseline | -0.06 (0.42) | 0.04 (0.22)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Regression, Linear; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.09 to 0.04]

9. Secondary Outcome: CGM-measured Hypoglycemia Events Per Week
Description: Change in number of CGM-measured hypoglycemia events per week (15 or more consecutive minutes <54 mg/dL) from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: events per week
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
events per week
  Baseline | 0.2 (0.3) | 0.1 (0.0)
  13 Weeks | 0.1 (0.2) | 0.1 (0.2)
  Change from Baseline | -0.1 (0.6) | 0.1 (0.3)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Regression, Linear; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.1 to 0.0]

10. Secondary Outcome: Coefficient of Variation
Description: Change in coefficient of variation mg/dL from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage SD of Mean
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
percentage SD of Mean
  Baseline | 28 (6) | 27 (5)
  13 Weeks | 30 (5) | 29 (5)
  Change from Baseline | 2 (5) | 2 (3)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Regression, Linear; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.5 to 1.2]

11. Other Pre Specified Outcome: HbA1c <7.0%
Description: Number of participants with HbA1c <7.0% at 13 weeks, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 214 | 104
Participants
  Baseline | 28 | 15
  13 Weeks | 78 | 28
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Test type: Superiority; Difference in percent of participants. = 12, 95% CI 2-sided [1 to 21] — Estimation represents the difference in percent of participants in each arm who achieved the outcome

12. Other Pre Specified Outcome: HbA1c <7.0% in Participants With Baseline HbA1c >7.5%
Description: Number of participants with HbA1c <7.0% at 13 weeks, in participants with baseline HbA1c >7.5%, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 214 | 104
Participants | 33 | 6
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Test type: Superiority; Difference in percent of participants. = 18, 95% CI 2-sided [2 to 32] — Estimation represents the difference in percent of participants in each arm who achieved the outcome

13. Other Pre Specified Outcome: HbA1c <7.5%
Description: Number of participants with HbA1c <7.5% at 13 weeks, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 214 | 104
Participants
  Baseline | 60 | 33
  13 Weeks | 132 | 44
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Test type: Superiority; Difference in percent of participants. = 23, 95% CI 2-sided [12 to 33] — Estimation represents the difference in percent of participants in each arm who achieved the outcome

14. Other Pre Specified Outcome: HbA1c Improvement From Baseline to 13 Weeks >0.5%
Description: Number of participants with HbA1c improvement from baseline to 13 weeks >0.5%, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 214 | 104
Participants | 123 | 31
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Test type: Superiority; Difference in percent of participants. = 25, 95% CI 2-sided [11 to 38] — Estimation represents the difference in percent of participants in each arm who achieved the outcome

15. Other Pre Specified Outcome: HbA1c Improvement From Baseline to 13 Weeks >1.0%
Description: Number of participants with HbA1c improvement from baseline to 13 weeks >1.0%, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 214 | 104
Participants | 81 | 14
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Test type: Superiority; Difference in percent of participants. = 22, 95% CI 2-sided [11 to 33] — Estimation represents the difference in percent of participants in each arm who achieved the outcome

16. Other Pre Specified Outcome: HbA1c Relative Improvement From Baseline to 13 Weeks >10%
Description: Number of participants with HbA1c relative improvement from baseline to 13 weeks >10%, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 214 | 104
Participants | 92 | 20
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Test type: Superiority; Difference in percent of participants. = 21, 95% CI 2-sided [10 to 32] — Estimation represents the difference in percent of participants in each arm who achieved the outcome

17. Other Pre Specified Outcome: HbA1c Improvement From Baseline to 13 Weeks >1.0% or HbA1c <7.0% at 13 Weeks
Description: Number of participants with HbA1c improvement from baseline to 13 weeks >1.0% or HbA1c <7.0% at 13 weeks, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 214 | 104
Participants | 130 | 42
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Test type: Superiority; Difference in percent of participants. = 21, 95% CI 2-sided [9 to 31] — Estimation represents the difference in percent of participants in each arm who achieved the outcome

18. Other Pre Specified Outcome: Time in Range 70-140 mg/dL
Description: Change in CGM percent time 70-140 mg/dL from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
percentage of time
  Baseline | 23 (18) | 23 (15)
  13 Weeks | 35 (15) | 25 (15)
  Change from Baseline | 12 (13) | 2 (11)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Median Difference (Net) = 10, 95% CI 2-sided [7 to 12]

19. Other Pre Specified Outcome: Area Over the Curve (70 mg/dL)
Description: CGM area over the curve (70 mg/dL), compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
mg*hr/dL
  Baseline | 0.07 (0.08) | 0.03 (0.03)
  13 Weeks | 0.04 (0.04) | 0.04 (0.04)
  Change from Baseline | -0.03 (0.16) | 0.02 (0.08)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Test type: Superiority; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.02 to 0.01]

20. Other Pre Specified Outcome: Low Blood Glucose Index
Description: Low blood glucose index (LBGI) by CGM with higher index indicating higher risk of hypoglycemia, compared between the intervention and control groups. LBGI ≤ 1.1 is associated with minimal risk of hypoglycemia, 1.1 < LBGI ≤ 2.5 is associated with a low risk of hypoglycemia, 2.5 < LBGI ≤ 5.0 is associated with a moderate risk of hypoglycemia, and LBGI > 5.0 is associated with high risk of hypoglycemia.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
units on a scale
  Baseline | 0.23 (0.24) | 0.12 (0.10)
  13 Weeks | 0.19 (0.15) | 0.17 (0.14)
  Change from Baseline | -0.04 (0.31) | 0.05 (0.17)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.07 to 0.01]

21. Other Pre Specified Outcome: Time >300 mg/dL
Description: Change in CGM percent time >300 mg/dL from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
percentage of time
  Baseline | 8.6 (9.4) | 6.4 (6.6)
  13 Weeks | 3.5 (3.6) | 6.8 (7.2)
  Change from Baseline | -5.1 (12.1) | 0.5 (8.5)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Mean Difference (Net) = -4.4, 95% CI 2-sided [-6.0 to -2.7]

22. Other Pre Specified Outcome: Area Under the Curve (180 mg/dL)
Description: CGM area under the curve (180 mg/dL), compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
mg*hr/dL
  Baseline | 34 (26) | 29 (21)
  13 Weeks | 19 (12) | 30 (21)
  Change from Baseline | -16 (27) | 1 (18)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Mean Difference (Net) = -14, 95% CI 2-sided [-18 to -10]

23. Other Pre Specified Outcome: High Blood Glucose Index
Description: High Blood Glucose Index (HBGI) by CGM, compared between the intervention and control groups., as a measure of Hyperglycemic Risk based on frequency and severity of hyperglycemic events. HBGI < 4.5 is associated with lower risk of hyperglycemia, 4.5 < HBGI < 9 is associated with a moderate risk of hyperglycemia and HBGI > 9 is associated with high risk of hyperglycemia.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
units on a scale
  Baseline | 12.6 (7.1) | 11.4 (5.6)
  13 Weeks | 8.1 (3.6) | 11.4 (5.8)
  Change from Baseline | -4.4 (6.8) | 0.0 (4.7)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Mean Difference (Net) = -3.9, 95% CI 2-sided [-5.2 to -2.7]

24. Other Pre Specified Outcome: Time in Range 70-180 mg/dL >70%
Description: Number of participants who achieved time in range 70-180 mg/dL >70%, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
Participants
  Baseline | 46 | 18
  13 Weeks | 81 | 23
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Test type: Superiority; Difference in percent of participants. = 16, 95% CI 2-sided [8 to 24] — Estimation represents the difference in percent of participants in each arm who achieved the outcome

25. Other Pre Specified Outcome: Time in Range 70-180 mg/dL Improvement From Baseline to 13 Weeks ≥5%
Description: Number of participants with time in range 70-180 mg/dL improvement from baseline to 13 weeks ≥5%, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
Participants | 149 | 43
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Test type: Superiority; Difference in percent of participants. = 26, 95% CI 2-sided [12 to 41] — Estimation represents the difference in percent of participants in each arm who achieved the outcome

26. Other Pre Specified Outcome: Time in Range 70-180 mg/dL Improvement From Baseline to 13 Weeks ≥10%
Description: Number of participants with time in range 70-180 mg/dL improvement from baseline to 13 weeks ≥10%, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Groups:
- AID Arm: t:slim X2 insulin pump with Control-IQ+ technology and Dexcom G6 CGM for 13 weeks.
Arm/Group | AID Arm | CGM Arm
Number analyzed (Participants) | 215 | 104
Participants | 122 | 20
Statistical Analysis 1: Comparison: AID Arm vs CGM Arm; Test type: Superiority; Difference in percent of participants. = 34, 95% CI 2-sided [21 to 45] — Estimation represents the difference in percent of participants in each arm who achieved the outcome

27. Other Pre Specified Outcome: Time <70 mg/dL <4%
Description: Number of participants with CGM time <70 mg/dL <4%, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
Participants
  Baseline | 207 | 104
  13 Weeks | 212 | 104

28. Other Pre Specified Outcome: Time <54 mg/dL <1%
Description: Number of participants with CGM time <54 mg/dL <1%, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
Participants
  Baseline | 205 | 103
  13 Weeks | 212 | 104

29. Other Pre Specified Outcome: Time in Range 70-180 mg/dL >70% and Time <54 mg/dL <1%
Description: Number of participants with time in range 70-180 mg/dL >70% and time <54 mg/dL <1%, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
Participants
  Baseline | 43 | 17
  13 Weeks | 80 | 23
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Test type: Superiority; Difference in percent of participants. = 15, 95% CI 2-sided [8 to 22] — Estimation represents the difference in percent of participants in each arm who achieved the outcome

30. Other Pre Specified Outcome: Total Insulin
Description: Total daily insulin delivery (units), compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: units/day
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
units/day
  Baseline | 95 (47) | 102 (50)
  13 Weeks | 87 (46) | 104 (56)
  Change from Baseline | -8 (38) | 2 (39)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Mean Difference (Net) = -10, 95% CI 2-sided [-20 to 0]

31. Other Pre Specified Outcome: Basal Insulin
Description: Percentage of insulin delivered as basal, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of units of insulin
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
percentage of units of insulin
  Baseline | 54.4 (16.1) | 52.6 (16.8)
  13 Weeks | 54.2 (11.9) | 54.1 (16.4)
  Change from Baseline | -0.2 (18.5) | 1.5 (17.8)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Mean Difference (Net) = -0.5, 95% CI 2-sided [-4.4 to 3.4]

32. Other Pre Specified Outcome: Weight
Description: Change in weight (kg) from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
kg
  Baseline | 100.5 (23.0) | 104.8 (25.5)
  13 Weeks | 103.1 (24.2) | 105.5 (24.5)
  Change from Baseline | 2.4 (4.4) | 0.9 (3.3)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Median Difference (Net) = 1.5, 95% CI 2-sided [0.5 to 2.5]

33. Other Pre Specified Outcome: Blood Pressure - Systolic
Description: Change in blood pressure (mm Hg) from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
mm Hg
  Baseline | 130 (17) | 128 (17)
  13 Weeks | 131 (17) | 129 (17)
  Change from Baseline | 1 (17) | 1 (15)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Mean Difference (Net) = 1.1, 95% CI 2-sided [-2.5 to 4.7]

34. Other Pre Specified Outcome: Blood Pressure - Diastolic
Description: Change in blood pressure (mm Hg) from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
mm Hg
  Baseline | 77 (11) | 77 (10)
  13 Weeks | 77 (11) | 78 (10)
  Change from Baseline | 0 (10) | 1 (9)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Mean Difference (Net) = -1.3, 95% CI 2-sided [-3.4 to 0.7]

35. Other Pre Specified Outcome: Lipid Levels - HDL
Description: Change in lipid levels (mg/dL) from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
mg/dL
  Baseline | 45.3 (11.9) | 44.9 (15.5)
  13 Weeks | 45.7 (12.3) | 43.7 (13.0)
  Change from Baseline | 0.7 (5.8) | -1.3 (7.1)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Median Difference (Net) = 2.1, 95% CI 2-sided [0.5 to 3.7]

36. Other Pre Specified Outcome: Lipid Levels - LDL
Description: Change in lipid levels (mg/dL) from baseline, compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
mg/dL
  Baseline | 75.6 (39.8) | 82.6 (40.6)
  13 Weeks | 77.9 (40.2) | 78.8 (36.6)
  Change from Baseline | 2.0 (27.1) | -5.3 (26.5)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Mean Difference (Net) = 4.9, 95% CI 2-sided [-1.4 to 11.1]

37. Other Pre Specified Outcome: Triglycerides
Description: Change in triglycerides (mg/dL), compared between the intervention and control groups
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
mg/dL
  Baseline | 164 (82) | 180 (96)
  13 Weeks | 157 (78) | 187 (108)
  Change from Baseline | -7 (77) | 7 (119)
Statistical Analysis 1: Comparison: Control-IQ+ AID vs CGM Arm; Adjusted Difference Between Groups; Test type: Superiority; Mean Difference (Net) = -20, 95% CI 2-sided [-45 to 4]

38. Other Pre Specified Outcome: Type 2 Diabetes Distress Assessment System (T2-DDAS Core and Source)
Description: Patient-reported outcome (PRO) measures from the Type 2 Diabetes Distress Assessment System (Core and Source) questionnaire, compared between the intervention and control groups. The T2-DDAS includes a Core measure that precisely characterizes the intensity of the emotional DD experience, and a set of Sources measures that identifies the key contributors or specific sources of distress. The seven Sources are: management demands, healthcare provider, hypoglycemia, long-term health, interpersonal issues, shame/stigma and healthcare access. Scoring for each question is on a scale of 1-5, with higher scores indicating more problems/distress. Scores are reported individually per domain area at baseline and 13 weeks.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
score on a scale
  Intensity Score - Baseline | 2.6 (1.1) | 2.6 (1.0)
  Intensity Score - 13 Weeks | 2.2 (1.0) | 2.4 (1.0)
  Hypoglycemia - Baseline | 2.0 (1.1) | 2.0 (1.1)
  Hypoglycemia - 13 Weeks | 1.9 (1.0) | 1.8 (1.0)
  Long-term health - Baseline | 2.6 (1.1) | 2.8 (1.2)
  Long-term health - 13 Weeks | 2.4 (1.1) | 2.5 (1.1)
  Healthcare provider - Baseline | 1.7 (0.9) | 1.7 (0.8)
  Healthcare provider - 13 Weeks | 1.5 (0.8) | 1.6 (0.8)
  Interpersonal issues - Baseline | 1.9 (1.0) | 1.9 (1.0)
  Interpersonal issues - 13 Weeks | 1.7 (0.9) | 1.7 (1.0)
  Shame/stigma - Baseline | 1.5 (0.8) | 1.5 (0.8)
  Shame/stigma - 13 Weeks | 1.4 (0.7) | 1.3 (0.8)
  Healthcare access - Baseline | 2.0 (0.9) | 2.1 (0.9)
  Healthcare access - 13 Weeks | 1.9 (0.9) | 2.0 (0.9)
  Management demands - Baseline | 2.6 (1.0) | 2.6 (1.1)
  Management demands - 13 Weeks | 2.3 (1.0) | 2.3 (1.0)

39. Other Pre Specified Outcome: DAWN Impact of Diabetes Profile (DIDP)
Description: Patient-reported outcome (PRO) measures from DAWN Impact of Diabetes Profile (DIDP) questionnaire, compared between the intervention and control groups. The DIDP provides a brief assessment of the perceived impact of diabetes on six key dimensions of life. Participants rate the impact of diabetes on each domain on a 7-point scale, with 1 being a very positive impact and 7 being a very negative impact. A converted percentage (0-100%) scale scores are reported. Lower scale scores indicate greater positive impact and higher scale scores indicate greater negative impact across global life dimensions.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 214 | 102
score on a scale
  Baseline | 59 (19) | 62 (15)
  13 Weeks | 59 (18) | 63 (15)

40. Other Pre Specified Outcome: Diabetes Impact and Satisfaction (DIDS) Scale
Description: Patient-reported outcome (PRO) measures from Diabetes Impact and Satisfaction (DIDS) Scale questionnaire, compared between the intervention and control groups. For the DIDS satisfaction score, scores range from 0-10 with higher scores indicating better outcome. For the DIDS impact score, scores range from 0-10 with lower scores indicating better outcome.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
score on a scale
  Device Satisfaction - Baseline | 6.7 (1.9) | 7.0 (1.9)
  Device Satisfaction - 13 Weeks | 8.2 (1.6) | 7.2 (1.8)
  Diabetes Impact - Baseline | 3.4 (1.7) | 3.3 (1.8)
  Diabetes Impact - 13 Weeks | 3.1 (1.7) | 3.4 (1.8)

41. Other Pre Specified Outcome: PROMIS Sleep-Related Impairment Questionnaire
Description: Patient-reported outcome (PRO) measures from PROMIS Sleep-Related Impairment questionnaire, compared between the intervention and control groups. The PROMIS Sleep-Related Impairment Questionnaire utilizes a T-score metric for scoring, with a mean of 50 and a standard deviation of 10. Higher T-scores indicate greater sleep-related impairment. The questionnaire uses a 5-point Likert scale (1=never to 5=always) for each item, and the responses are summed to calculate a total raw score. This raw score is then converted to a T-score using a lookup table provided in the scoring manual.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 214 | 104
score on a scale
  Baseline | 22.4 (7.3) | 22.0 (7.1)
  13 Weeks | 19.6 (6.9) | 21.8 (7.4)

42. Other Pre Specified Outcome: System Usability Scale (SUS)
Description: Patient-reported outcome (PRO) measures from System Usability Scale (SUS) questionnaire, compared between the intervention and control groups. 10 items rated on 5-point Likert scale (1=Strongly Disagree, 5=Strongly Agree). Total score is on a 100 point scale (0 - 100), with higher scores indicating greater usability.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
score on a scale
  Baseline | 69 (18) | 70 (18)
  13 Weeks | 75 (19) | 73 (17)

43. Other Pre Specified Outcome: Hypoglycemia Fear Survey II
Description: Patient-reported outcome (PRO) measures from Hypoglycemia Fear Survey II Behavior and Worry Scores, compared between the intervention and control groups. The HFS-II consists of 33 items, which are organized into two subscales: HFS-B (Behavior): A 15 item subscale that focuses on behaviors to avoid hypoglycemia, and HFS-W (Worry): a 18 item subscale that focuses on worries about hypoglycemia and its consequences. The HFS-II subscale scores range from 0-60 and 0-72 for the HFS-B and HFS-W, respectively. Higher scores indicate higher fear of hypoglycemia.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
score on a scale
  Behavior - Baseline | 27 (18) | 30 (18)
  Behavior - 13 Weeks | 26 (17) | 28 (17)
  Worry - Baseline | 22 (23) | 22 (19)
  Worry - 13 Weeks | 19 (20) | 21 (21)

44. Other Pre Specified Outcome: EQ5D-5L
Description: Patient-reported outcome (PRO) measures from EQ5D-5L questionnaire, compared between the intervention and control groups, showing EQ-Index Scores. The EQ5D utility index consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response categories, from which a single EQ-5D index score can be calculated ranging from 0 (worst imaginable health) to 1 (best imaginable health) on which participants have to indicate their current health.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control-IQ+ AID | CGM Arm
Number analyzed (Participants) | 215 | 104
score on a scale
  EQ-Index - Baseline | 0.76 (0.22) | 0.75 (0.27)
  EQ-Index - 13 Weeks | 0.77 (0.24) | 0.74 (0.29)

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | Control-IQ+ AID | CGM Arm
All-Cause Mortality (participants affected / at risk) | 0/215 | 1/104
Serious Adverse Events (participants affected / at risk) | 17/215 | 7/104
Other Adverse Events (participants affected / at risk) | 60/215 | 18/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control-IQ+ AID (N=215) | CGM Arm (N=104)
Severe Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Endocrine disorders) | 0 (0) | 0 (0)
Hyperosmolar hyperglycemic syndrome (Endocrine disorders) | 0 (0) | 0 (0)
Back surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast ductal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Chest pressure (Cardiac disorders) | 1 (1) | 0 (0)
Congestive heart failure (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Vascular disorders) | 0 (0) | 1 (1)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Foot infection (Infections and infestations) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1)
Hip fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Infection (chronic) of amputation stump (Infections and infestations) | 1 (1) | 0 (0)
Knee surgery NOS (Surgical and medical procedures) | 1 (1) | 0 (0)
Multinodular goiter (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Other specified adverse effect, not elsewhere classified (General disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Fatal) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Total knee replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Unstable angina (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vitreous hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control-IQ+ AID (N=215) | CGM Arm (N=104)
Hyperglycemia with or without ketosis related to study device (Endocrine disorders) | 13 (20) | 0 (0)
Hyperglycemia with or without ketosis not related to study device (Endocrine disorders) | 1 (1) | 2 (2)
Non-severe hypoglycemia (Endocrine disorders) | 9 (10) | 2 (2)
Other reportable adverse events (General disorders) | 37 (56) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/32/NCT05785832/Prot_001.pdf
  • Statistical Analysis Plan (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT05785832/SAP_002.pdf